

# **Non-Interventional Study (NIS) Protocol**

| Document Number: | c37262534-01 |
|---|---|
| BI Study Number: | 1237-0113 |
| BI Investigational Product(s): | Stiolto Respimat (Tiotropium Bromide/Olodaterol) |
| Title: | Health Care Resource Utilization, Cost and Other Outcomes of<br>Patients Diagnosed with COPD Initiating Tiotropium<br>Bromide/Olodaterol versus Fluticasone<br>Furoate/Umeclidinium/Vilanterol |
| Brief lay title: | Outcomes among COPD patients initiating TIO/OLO vs FF/UMEC/VI |
| Protocol version identifier: | Version 1.0 |
| Date of last version of protocol: | 04 May 2021 |
| PASS: | No |
| EU PAS register number: | Study not registered |
| Active substance: | Tiotropium Bromide/Olodaterol |
| Medicinal product: | Stiolto Respimat (Tiotropium Bromide/Olodaterol) |
| Product reference: | NA |
| Procedure number: | NA |
| Marketing authorisation holder(s): | Boehringer Ingelheim |
| Joint PASS: | NA |
| Research question and objectives: | The purpose of this study is to estimate disease-related and all-cause burden and clinical outcomes of interest following initiation of COPE maintenance therapy with TIO/OLO or FF/UMEC/VI. |
| L | ı |

NIS Protocol 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Country(-ies) of study: | United States |
|---|---|
| Author: | Boehringer Ingelheim: |
| Marketing authorisation holder(s): | NA |
| In case of PASS, add: MAH contact person: | NA |
| In case of PASS, add: <eu-qppv:></eu-qppv:> | NA |
| In case of PASS, add: <signature eu-="" of="" qppv:=""></signature> | NA |
| Date: | 04 May 2021 |
| Proprietary confidential information © 2022 Boehringer Ingelheim Group of companies. All rights reserved. This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission | |

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 1. **TABLE OF CONTENTS**

| TITLE PA | AGE | 1 |
|----------|-------------------------------------------------|----|
| 1. TAB | LE OF CONTENTS | 3 |
| 2. LIST | OF ABBREVIATIONS | 5 |
| 3. RESI | PONSIBLE PARTIES | 6 |
| 4. ABS | TRACT | 7 |
| 5. AME | ENDMENTS AND UPDATES | 11 |
| 6. MILI | ESTONES | 12 |
| 7. RAT | IONALE AND BACKGROUND | 13 |
| 8. RESI | EARCH QUESTION AND OBJECTIVES | 15 |
| 9. RESI | EARCH METHODS | 16 |
| 9.1 | STUDY DESIGN | 16 |
| 9.2 | SETTING | 17 |
| 9.2.1 | Observation period | 17 |
| 9.2.2 | Observation period – secondary objective | 19 |
| 9.2.3 | Study sites | 19 |
| 9.2.4 | Study population | 19 |
| 9.2.4 | .1 Patient Identification – Eosinophil Subgroup | 20 |
| 9.2.5 | Study visits | 21 |
| 9.2.6 | Study discontinuation | 21 |
| 9.3 | VARIABLES | 21 |
| 9.3.1 | Exposures | 21 |
| 9.3.2 | Outcomes | 21 |
| 9.3.2 | .1 Primary outcomes | 21 |
| 9.3.2 | .2 Secondary outcomes | 25 |
| 9.3.3 | Covariates | 26 |
| 9.3.3 | .1 Clinical Characteristics | 26 |
| 9.3.3 | .2 Patient Characteristics | 29 |
| 9.4 | DATA SOURCES | 30 |
| 9.4.1 | Database | 30 |
| 9.4.2 | Laboratory Results | 31 |
| 9.5 | STUDY SIZE | 31 |

**NIS Protocol** 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| 9.6 | DATA MANAGEMENT | 31 |
|------------------|---------------------------------------------------|-----|
| 9.7 | DATA ANALYSIS | 32 |
| 9.7.1 | Comparison of TIO/OLO Initiators | 32 |
| 9.7.2 | Main analysis | 32 |
| 9.7.3 | Primary Objectives | 33 |
| 9.7.3.1 | Descriptive Analysis | 33 |
| 9.7.3.2 | Kaplan Meier Analysis | 34 |
| 9.7.3.3 | Number Needed to Treat | 34 |
| 9.7.3.4 | Multivariable Analysis (Optional) | 34 |
| 9.7.4 | Secondary Objective. | 35 |
| 9.7.4.1 | COPD Readmission CMS Definition | 35 |
| 9.8 | LIMITATIONS OF THE RESEARCH METHODS | 36 |
| 9.9 | OTHER ASPECTS | 37 |
| 9.9.1 | Data quality assurance | 37 |
| 9.9.2 | Study records | 37 |
| 9.9.2.1 | Source documents | 37 |
| 10. | PROTECTION OF HUMAN SUBJECTS | 38 |
| 10.1<br>CONSENT | STUDY APPROVAL, PATIENT INFORMATION, AND INFORMED | 38 |
| 10.2 | STATEMENT OF CONFIDENTIALITY | |
| 11.<br>REACTION | MANAGEMENT AND REPORTING OF ADVERSE EVENTS/ADVE | |
| 11.1<br>AND REPO | ADVERSE EVENT AND SERIOUS ADVERSE EVENT COLLECTIO | |
| 12.<br>RESULTS | PLANS FOR DISSEMINATING AND COMMUNICATING STUDY | 40 |
| 13. | REFERENCES | 41 |
| 13.1 | PUBLISHED REFERENCES | 41 |
| ANNEX 1. | LIST OF STAND-ALONE DOCUMENTS | 43 |
| ANNEX 2. | ENCEPP CHECKLIST FOR STUDY PROTOCOLS | 44 |
| ANNEX 3. | ADDITIONAL INFORMATION | 45 |
| ANNEY 4 | REVIEWERS AND APPROVAL SIGNATURES | 252 |

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 2. LIST OF ABBREVIATIONS

CI Confidence Intervals

**CMS** Centers for Medicare and Medicaid Services **COPD** Chronic Obstructive Pulmonary Disease

CPI Consumer Price Index

**CPT** Current Procedural Terminology

**Emergency Department** ED

**EPO Exclusive Provider Organization** 

**Emergency Room** ER

Food and Drug Administration **FDA** Fixed Dose Combination **FDC** 

Global Initiative for Chronic Obstructive Lung Disease **GOLD** 

**HCFA** Health Care Financing Administration Healthcare Common Procedure Coding **HCPCS** Health Care Resource Utilization HCRU

**HIPAA** Health Insurance Portability and Accountability Act

**HMO** Health Maintenance Organization Health Professional Shortage Areas **HPSA** 

International Statistical Classification of Diseases and Related Health **ICD** 

**Problems** 

**ICS** Inhaled Corticosteroid

**IMPACT** InforMing the Pathway of COPD Treatment

Kaplan-Meier KM

Long-acting ß-agonist LABA Long-acting Antimuscarinic LAMA Medicare Advantage Part D MAPD

Number Needed to Treat **NNT** 

Oral Corticosteroid **OCS** Database D

POS Point of Service

PPO Preferred Provider Organization **PSM Propensity Score Matching** SABA Short-acting \( \mathbb{B}\)-agonist

**Short-acting Anticholinergics SAMA** 

Tiotropium/Olodaterol TIO/OLO

Triple Therapy TT Uniform Billing UB Umeclidinium **UMEC United States** US VI Vilanterol

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### **3. RESPONSIBLE PARTIES**

**NIS Protocol** 



001-

 **NIS Protocol** Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## **ABSTRACT**

| Name of company: | | | |
|---|---|---|---|
| Boehringer Ingelheim | | | |
| Name of finished medicinal product: Stiolto Respimat | | | |
| Name of active ingr<br>Tiotropium Bromide | | | |
| Protocol date: | Study<br>number: | Version/Revision: | Version/Revision date: |
| 04 May 2021 | 1237-0113 | 1.0 | NA |
| Title of study: | Diagnosed with | ource Utilization, Cost and Oth<br>COPD Initiating Tiotropium Br<br>pate/Umeclidinium/Vilanterol | |
| Rationale and background: | The Global Initiative for Chronic Obstructive Lung Disease (GOLD) 2020 report recommends dual therapy with long-acting muscarinic antagonists (LAMAs) plus long-acting beta <sub>2</sub> agonists (LABAs) for patients with chronic obstructive pulmonary disease (COPD) who have persistent symptoms and/or exacerbations on LAMA or LABA monotherapy. Consideration of escalation to triple therapy (TT; LAMA+LABA+inhaled corticosteroids [ICS]) is recommended in case of further exacerbation and after assessing the risks/benefits, including the increased risk of pneumonia with ICS treatment. A blood eosinophil count >300 cells/μL and exacerbation history together can be used to identify patients with the greatest likelihood of treatment benefit with ICS. Despite these recommendations, evidence suggests TT is over-prescribed across all COPD severities, including those at low exacerbation risk. This deviation from GOLD recommendations may have economic and clinical consequences. | | |
| | and LAMA/LAE study only one tr - compared FDC Trelegy Ellipta) [UMEC/VI; An exacerbation rate cause mortality of the study | tiple Phase III randomized clinical trials comparing FDC TT aBA are currently available. However, for the purposes of this trial - InforMing the PAthway of COPD Treatment (IMPACT) C fluticasone furoate/umeclidinium/vilanterol (FF/UMEC/VI; a) and LAMA/LABA (specifically umeclidinium/vilanterol Anoro Ellipta]). The study found significantly lower ates, higher pneumonia rates [R18-1532], and reduction in allorisk [R21-4089] for FF/UMEC/VI. | |
| Research question and objectives: | The purpose of this study is to estimate disease-related and all-cause burden and clinical outcomes of interest following initiation of COPD maintenance therapy with TIO/OLO or FF/UMEC/VI. | | |

Stiolto vs Trelegy V1.0 04 May 2021 MCS-90-118\_RD-23 (1.0) / Saved on: 25 Nov 2019 001-

001-

NIS Protocol 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### Study design:

This will be a retrospective study of commercial and MAPD beneficiaries, using administrative claims data for the period of 01 January 2013 through 31 December 2019. This study will include patients diagnosed with COPD who initiated treatment with TIO/OLO or FF/UMEC/VI between 01 June 2015 and 30 November 2019. Patients will be assigned to one of the following mutually exclusive study cohorts based on the index pharmacy claim: TIO/OLO or FF/UMEC/VI. Stratified propensity score matching (PSM), using an exact match on some variables and a propensity score match on the others, will be used to control for possible confounding of the association between the outcomes (e.g., health care resource utilization) and treatment with TIO/OLO or FF/UMEC/VI.

#### Population:

#### **Inclusion Criteria**

- ≥30 consecutive days with TIO/OLO or FF/UMEC/VI initiated during the patient identification period of 01 June 2015 to 30 November 2019. The *index date* will be the date of the TIO/OLO or FF/UMEC/VI pharmacy claim that starts the ≥30 consecutive days with the medication.
- ≥1 facility claim with a diagnosis of COPD in the primary position or ≥2 professional claims with a diagnosis code for COPD (Annex 3) in any position on separate dates of service during the study period
- $\geq$ 40 years of age as of the year of the index date
- Continuous enrollment with medical and pharmacy coverage for 12 months prior to and including the index date (baseline period)
- Continuous enrollment with medical and pharmacy coverage for ≥30 days following the index date and without discontinuation of the index medication or switch to a non-index regimen (follow-up period); discontinuation and switch are defined in Section 9.2.1.

#### **Exclusion Criteria**

- ≥2 medical claims with a diagnosis code for asthma, cystic fibrosis, lung cancer, or interstitial lung disease (Annex 3) in any position on separate dates of service during the baseline period
- Pharmacy claims for both TIO/OLO and FF/UMEC/VI on the index date
- A pharmacy claim for any non-index COPD maintenance medication on the index date, defined as: LAMA monotherapy; LABA monotherapy; ICS monotherapy; FDC ICS/LABA, or FDC LAMA/LABA (Annex 3)
- Free or fixed dose LAMA+LABA maintenance therapy defined as ≥7 consecutive days of overlapping days' supply with a LAMA and LABA during a 6-month pre-index period, excluding the index date (Annex 3)

c37262534-01

NIS Protocol 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Flags will be created to identify patients excluded for baseline LAMA/LABA use overall and specifically for each FDC LAMA/LABA medication Free or fixed dose TT defined as ≥7 consecutive days of overlapping days' supply with an ICS, LABA, and LAMA during a 6-month preindex period, excluding the index date (Annex 3) ≥1 medical claim with a procedure code for lung volume reduction during the study period (Annex 3) Unknown age, gender, or business line, or unknown/other geographic region The exclusion criteria for previous medication use was relaxed to  $\geq 7$ consecutive days of overlapping days' supply rather than ≥1 day of overlapping days' supply based on the number of patients excluded in the attrition table. This decision was made after reviewing the attrition tables using the two criteria and before any baseline or follow-up analyses were completed. Study inclusion and exclusion criteria will be finalized during review of the patient attrition table, and prior to any baseline or follow-up analyses. Variables: Patients will be assigned to one of the following mutually exclusive study cohorts based on the index pharmacy claim: TIO/OLO or FF/UMEC/VI. COPD and/or pneumonia-related costs and HRU COPD-related costs and HRU Pneumonia-related costs and HRU All-cause costs and HRU COPD or pneumonia-attributable costs and HRU COPD exacerbations Pneumonia diagnoses Pneumonia-related hospitalization COPD exacerbation and/or pneumonia diagnosis **Baseline characteristics** Clinical and demographic characteristics HRU Costs The Database ( D), is fully de-identified and HIPAA **Data sources:** compliant, and comprised of medical and pharmacy claims data (including linked enrollment information) from 1993 to present on more than 73 million lives. Using claims data for commercial and Medicare Advantage health plan **Study size:** 

Stiolto vs Trelegy V1.0 04 May

enrollees we identified 5,717 and 17,733 patients who initiated treatment

**NIS Protocol** 

c37262534-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| | with TIO/OLO or FF/UMEC/VI, respectively, between 01 January 2018 and 31 July 2019. These patients had 12-months of baseline and ≥30 days of follow-up continuous enrollment with both medical and pharmacy coverage. This count is for informational purposes only and may not represent the actual number of patients to be utilized in the study. Application of other inclusion and exclusion criteria required for this study or other factors may reduce the sample size. |
|---|---|
| Data analysis: | Baseline categorical variables will be presented as numbers and percentages and baseline continuous variables will be presented as means, standard deviations, medians, and interquartile ranges. Follow-up variables will be presented as population annualized averages to account for the variable follow-up duration (minimum 1 month, maximum 12 months). Population annualized averages will be calculated as ([sum of all utilization or cost for all individuals during the follow-up period]/[sum of all follow-up time in days for all individuals])*365. Wald 95% confidence intervals (CI) will be provided for annualized population averages using the Taylor expansion to estimate the standard error. The numerator and denominator of the population annualized average equation and the 95% CI will be presented. Appropriate tests comparing the TIO/OLO cohort and the FF/UMEC/VI cohort (e.g., standardized differences, McNemar's tests, paired t-tests, sign tests) will be used based on the distribution of the measure. |
| Milestones: | Final report planned: March 2022 |

001-

c37262534-01

001-

**NIS Protocol**  Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### **AMENDMENTS AND UPDATES 5.**

None

c37262534-01

 **NIS Protocol** Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### **MILESTONES 6.**

| Milestone | Planned Date |
|--------------------------------|--------------|
| Final report of study results: | March 2022 |

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 7. RATIONALE AND BACKGROUND

**NIS Protocol** 

The Global Initiative for Chronic Obstructive Lung Disease (GOLD) 2020 report recommends dual therapy with long-acting muscarinic antagonists (LAMAs) plus long-acting beta<sub>2</sub> agonists (LABAs) for patients with chronic obstructive pulmonary disease (COPD) who have persistent symptoms and/or exacerbations on LAMA or LABA monotherapy. Consideration of escalation to triple therapy (TT; LAMA+LABA+inhaled corticosteroids [ICS]) is recommended in case of further exacerbation and after assessing the risks/benefits, including the increased risk of pneumonia with ICS treatment. A blood eosinophil count >300 cells/μL and exacerbation history together can be used to identify patients with the greatest likelihood of treatment benefit with ICS. Despite these recommendations, evidence suggests TT is over-prescribed across all COPD severities, including those at low exacerbation risk. This deviation from GOLD recommendations may have economic and clinical consequences.

A recently completed retrospective observational claims analysis of COPD patients enrolled in a Medicare-Advantage with Part D (MAPD) coverage plan, compared on-treatment COPD related healthcare cost and resource utilization (HCRU) among patients initiating tiotropium/olodaterol (TIO/OLO) vs. TT. Findings using propensity score matched cohorts included 41% (\$7,041) lower annualized cost per patient for TIO/OLO vs. TT (\$10,094 vs. \$17,135, P<.001) [P20-06571].

A *post-hoc* analysis of the same population examined outcomes for TIO/OLO and TT cohorts by stratifying on maintenance naïve status (no baseline COPD maintenance medications) and baseline exacerbation history (0 exacerbations, 1 moderate and no severe exacerbations, and ≥2 moderate or ≥1 severe exacerbations) and then matching on patient characteristics. Across these various subgroups, post-propensity score match, COPD-related annual costs for TIO/OLO versus TT were found to be significantly lower, with the greatest differences among the maintenance naïve and no exacerbation history subgroups, with 47% (\$8,018) and 53% (\$8,478) lower annual costs per patient, respectively. Cost differences in both subgroups were driven by COPD-related medical costs with 57% and 60% contribution, respectively, towards the observed total difference. Composite COPD/pneumonia related costs for TIO/OLO were similarly lower in the maintenance naïve (47% [\$9,548]) and no exacerbation history subgroups (56% [\$10,274]) compared to TT.

The same analysis also examined exacerbation and pneumonia diagnosis outcomes. After adjusting for treatment and additional covariates, the risk for a severe exacerbation was approximately 57% lower, for TIO/OLO patients with no exacerbation history compared to TT patients (P=0.002). The risk for pneumonia or acute bronchitis/bronchiolitis was approximately 34% lower among the TIO/OLO cohort with no exacerbation history compared to the TT cohort (P=0.018). However, the generalizability of these findings to contemporary TT initiators is limited since the TT cohort was predominantly composed of free-dose TT combinations. Only 1% involved fixed-dose combination (FDC) TT owing to the study end date.

**NIS Protocol** 

c37262534-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Data from multiple Phase III randomized clinical trials comparing FDC TT and LAMA/LABA are currently available. However, for the purposes of this study only one trial -InforMing the PAthway of COPD Treatment (IMPACT) - compared FDC fluticasone furoate/umeclidinium/vilanterol (FF/UMEC/VI; Trelegy Ellipta) and LAMA/LABA (specifically umeclidinium/vilanterol [UMEC/VI; Anoro Ellipta]). The study found significantly lower exacerbation rates, higher pneumonia rates [R18-1532], and reduction in all-cause mortality risk [R21-4089] for FF/UMEC/VI. Additionally, a recently completed post-hoc, within trial economic analysis of this trial data found that FF/UMEC/VI resulted in lower 1-year on-treatment COPD exacerbation-related costs that were attributable to the lower exacerbation events for FDC TT rates from the trial [R21-4088]. However, both the trial and this post-hoc analysis have a few significant limitations in design and generalizability. Primarily, the trial itself involved a predominately severe COPD patient population of frequent exacerbators or GOLD C/D patients (70% were GOLD Group D and 74% had at least 2 moderate and/or 1 severe exacerbation in the year preceding the trial) and is not representative of the general COPD population. And the post-hoc analysis was further limited since it did not account for costs of maintenance treatment and pneumonia events, which may have offset the cost savings observed for FF/UMEC/VI.

Following the approval of FF/UMEC/VI FDC TT in late 2017 for the long-term maintenance treatment of COPD, this study attempts to fill the existing real-world evidence gap by comparing TIO/OLO vs. FF/UMEC/VI. We aim to understand the clinical and economic implications of prescribing FDC TT vs. TIO/OLO in clinical practice.

NIS Protocol 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 8. RESEARCH QUESTION AND OBJECTIVES

The purpose of this study is to estimate disease-related and all-cause burden and clinical outcomes of interest following initiation of COPD maintenance therapy with TIO/OLO or FF/UMEC/VI.

The specific primary objectives for this project are:

- To compare disease related and all-cause HCRU among patients newly treated with TIO/OLO compared with patients newly treated with FF/UMEC/VI
- To compare disease-related and all-cause medical and total (medical & pharmacy) health care costs among patients newly treated with TIO/OLO compared with patients newly treated with FF/UMEC/VI
- To compare pneumonia outcomes among patients newly treated with TIO/OLO compared with patients newly treated with FF/UMEC/VI
- To compare COPD exacerbations following initiation of TIO/OLO or FF/UMEC/VI

The specific secondary objective for this project is:

• To compare 30-day all-cause hospital readmissions following initiation of TIO/OLO or FF/UMEC/VI

The study objectives will be assessed within each of the following populations of TIO/OLO and FF/UMEC/VI initiators:

- Overall population of initiators (i.e., initiators who meet study selection criteria)
- Maintenance naïve (patients with no baseline maintenance medication [no free or fixed dose combination (FDC) LAMA, LABA, or ICS])
- No exacerbation (patients with no baseline exacerbation)
- No exacerbation or 1 exacerbation not leading to hospitalization (i.e., baseline GOLD A/B)
- ≥2 exacerbations not leading to hospitalization or ≥1 exacerbation leading to hospitalization [i.e., baseline GOLD C/D])

Additionally, HCRU, costs, COPD exacerbations, and pneumonia outcomes following initiation of TIO/OLO or FF/UMEC/VI will be assessed among subgroups of patients with ≥1 eosinophil lab in the following groups:

- Baseline blood eosinophil count ≤300 cells/μL
- Baseline blood eosinophil count >300 cells/µL

NIS Protocol 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 9. RESEARCH METHODS

#### 9.1 STUDY DESIGN

This will be a retrospective study of commercial and MAPD beneficiaries, using administrative claims data for the period of 01 January 2013 through 31 December 2019. Due to the COVID-19 pandemic, no data from 2020 will be included in this analysis. Medical claims are approximately 95% complete (fully adjudicated) approximately four to six months following the date of service. Pharmacy claims are complete (fully adjudicated) in the database approximately six weeks following the date of service. Laboratory results are typically added to the database within three to six months of administration of the test.

This study will include commercial and MAPD health plan members diagnosed with COPD who initiated treatment with TIO/OLO or FF/UMEC/VI between 01 June 2015 and 30 November 2019. The start of the patient identification period is based on the Food and Drug Administration (FDA) approval date of 21 May 2015 for use of TIO/OLO (i.e., Stiolto) for treatment of COPD, and may be moved later (e.g., 01 August 2015) based on uptake of TIO/OLO within the

Ideally the patient identification period would only include the time period when both TIO/OLO and FF/UMEC/VI were approved for treatment of COPD. However, FF/UMEC/VI was FDA-approved for the treatment of COPD on 18 September 2017, and starting patient identification in January 2018 (to allow for uptake of FF/UMEC/VI in the D), would substantially reduce the number of TIO/OLO patients identified the study. Since meaningful effect sizes for the study comparisons currently are unknown, and the primary analysis focuses on key subgroups of initiators (e.g., maintenance naïve), the patient identification period will begin at TIO/OLO approval.

TIO/OLO initiators with index dates before and after the FF/UMEC/VI approval data will be compared on a list of a priori baseline characteristics. The analytic plan, including the threshold for deciding if the TIO/OLO initiators are similar before and after FF/UMEC/VI approval is outlined in <a href="Section 9.7.1">Section 9.7.1</a>

Stratified propensity score matching (PSM), using an exact match on some variables and a propensity score match on the others, will be used to control for possible confounding of the association between the outcomes (e.g., health care resource utilization) and treatment with TIO/OLO or FF/UMEC/VI. This methodology has been widely used in observational studies for causal inference ever since it was introduced by Rosenbaum and Rubin.4 Depending on pre-match cohort sizes, patients will be matched in a 1:1 or 1:2 ratio of TIO/OLO to FF/UMEC/VI. Patients not matched will be excluded from the post-match analysis.

Covariates for the stratified match may include:

- Baseline exacerbation (number of severe and number of moderate exacerbations; yes/no)
- Bronchodilator naïve status (naïve to LAMA and LABA)

c37262534-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Potential covariates for the logistic regression model include:

• Index year, seasonality

**NIS Protocol** 

- Patient demographics: age, gender, geographic region
- Baseline medication use: controller and rescue
- Baseline comorbidity burden (e.g., Quan-Charlson Comorbidity Score without COPD)
- Baseline healthcare utilization: all-cause, COPD-related, pneumonia-related
- Baseline healthcare costs: all-cause, COPD-related, pneumonia-related

The final list of variables to be included in the propensity score modeling will be determined following review of the pre-matching descriptive analysis of patient characteristics and other baseline measures.

The success of the matching procedure will be evaluated by comparing the characteristics included in the propensity score model between cohorts using standardized differences and other measures. Modifications may be made to the propensity score modeling procedure to increase sample size or improve balance between the cohorts. A standardized difference of  $\leq 10\%$  for a measure will be considered as an acceptable threshold for balance between the treatment cohorts.

Statistical tests between cohorts will include variance adjustments for the clustering due to matching.

A separate stratified PSM will be conducted among the subgroup of TIO/OLO and FF/UMEC/VI patients with baseline eosinophil laboratory results. The methodology applied to the overall sample will be replicated for this subgroup analysis. If the numbers allow, patients in the subgroup analysis will be hard matched on baseline exacerbation history, baseline bronchodilator naïve status, and baseline eosinophil level (eosinophil >300 cells/ $\mu$ L) or eosinophil  $\leq$ 300 cells/ $\mu$ L) and propensity score matched on other baseline variables.

As an alternative approach, inverse probability of treatment weighting (IPTW) may be conducted in lieu of PSM.

#### 9.2 SETTING

#### 9.2.1 Observation period

Patients will be required to be continuously enrolled in the health plan for a minimum of 13 months. A schematic of the observation period is presented in <u>Figure 1</u>

- **Baseline period:** The 12 months prior to and including the index date (index date—364 through index date) will be used to assess baseline patient and clinical characteristics. The index pharmacy claims will be excluded from the baseline period and included in the follow-up period.
- **Follow-up period:** The variable period starting on the day after the index date, with a minimum of 30-days duration (index date+1 through index date+30) up to a

**NIS Protocol** 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

maximum of 12 months duration (index date+1 through index date+365) will be used to assess HCRU, costs, exacerbation and pneumonia outcomes. Patients will be censored at the earliest of the following: discontinuation of the index medication, switch to a non-index regimen, disenrollment from the health plan, 12-months following the index date, or the end of the study period.

- <u>Discontinuation</u> will be defined as a gap in therapy of ≥60 days following the runout of days supply (discontinuation date = runout prior to the gap). Because the discontinuation status of patients whose runout of index medication occurs <60 days before the end of their observation time is unobservable, patients with <60 days of observation time following the runout of their last index prescription claim will be flagged as censored, and their observation period will end on the runout date.
- <u>Switch</u> will be defined as a pharmacy fill for ≥30 consecutive days of a non-index ICS-, LABA-, or LAMA-containing medication (switch date = first date of the new treatment regimen).

The distribution of follow-up time will be compared between the study cohorts. If there is a difference of more than one month of follow-up time between the cohorts, one or more of the following options may be utilized: for binary outcomes, a Kaplan-Meier analyses restricted to when both cohorts have follow-up time; for continuous outcomes, censoring the follow-up period of the cohort with longer follow-up such that the analysis is restricted to when both cohorts have follow-up time; for each matched pair (TIO/OLO and FF/UMEC/VI), use the minimum of follow-up time for the pair; include follow-up time in the propensity score match; or an alternative approach.

Figure 1 Observation Period for HCRU and Cost, COPD Exacerbation, and Pneumonia Outcomes



Stiolto vs Trelegy V1.0 04 May

001-

001-

NIS Protocol 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 9.2.2 Observation period – secondary objective

A hospitalization-level analysis will be used to examine 30-day all-cause hospital readmission after a COPD-related hospitalization while on the index regimens of interest. To be included in the readmission analysis, patients must meet the study selection criteria outlined in Section 9.2.4. plus have ≥1 eligible COPD-related hospitalization in the follow-up period with at least 30 days of continuous enrollment after discharge, unless readmission and death occur within 30 days of hospital discharge. Among patients who meet the study selection criteria, 30-day all-cause readmission following a COPD-related hospitalization while on the index regimens will be performed. Patients may contribute zero, one, or more than one observation depending on the number of COPD-related inpatient visits observed during follow-up. Each COPD-related hospitalization will be required to have at least 30 days of enrollment after the discharge date to be included in the analysis, unless readmission and death occur within 30 days of hospital discharge. Hospitalization discharge dates that occur within 30 days of the study end date will not be included because the readmission status is unobservable.

### 9.2.3 Study sites

The Database (D), is fully de-identified and HIPAA compliant, and comprised of medical and pharmacy claims data (including linked enrollment information) from 1993 to present on more than 73 million lives.

### 9.2.4 Study population

Patients will be assigned to one of the following mutually exclusive study cohorts based on the index pharmacy claim: TIO/OLO or FF/UMEC/VI.

#### **Inclusion Criteria**

- ≥30 consecutive days with TIO/OLO or FF/UMEC/VI initiated during the patient identification period of 01 June 2015 to 30 November 2019. The *index date* will be the date of the TIO/OLO or FF/UMEC/VI pharmacy claim that starts the ≥30 consecutive days with the medication.
- ≥1 facility claim with a diagnosis of COPD in the primary position or ≥2 professional claims with a diagnosis code for COPD (Annex 3) in any position on separate dates of service during the study period
- $\geq$ 40 years of age as of the year of the index date
- Continuous enrollment with medical and pharmacy coverage for 12 months prior to and including the index date (baseline period)
- Continuous enrollment with medical and pharmacy coverage for ≥30 days following the index date and without discontinuation of the index medication or switch to a non-index regimen (follow-up period); discontinuation and switch are defined in <u>Section</u> 9.2.1.

panies c37262534-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### **Exclusion Criteria**

NIS Protocol

- ≥2 medical claims with a diagnosis code for asthma, cystic fibrosis, lung cancer, or interstitial lung disease (<u>Annex 3</u>) in any position on separate dates of service during the baseline period
- Pharmacy claims for both TIO/OLO and FF/UMEC/VI on the index date
- A pharmacy claim for any *non-index* COPD maintenance medication on the index date, defined as: LAMA monotherapy; LABA monotherapy; ICS monotherapy; FDC ICS/LABA, or FDC LAMA/LABA (Annex 3)
- Free or fixed dose LAMA+LABA maintenance therapy defined as ≥7 consecutive days of overlapping days' supply with a LAMA and LABA during a 6-month preindex period, excluding the index date (Annex 3)
  - Flags will be created to identify patients excluded for baseline LAMA/LABA use overall and specifically for each FDC LAMA/LABA medication
- Free or fixed dose TT defined as ≥7 consecutive days of overlapping days' supply
  with an ICS, LABA, and LAMA during a 6-month pre-index period, excluding the
  index date (Annex 3)
- ≥1 medical claim with a procedure code for lung volume reduction during the study period (Annex 3)
- Unknown age, gender, or business line, or unknown/other geographic region

The exclusion criteria for previous medication use was relaxed to  $\geq 7$  consecutive days of overlapping days' supply rather than  $\geq 1$  day of overlapping days' supply based on the number of patients excluded in the attrition table. This decision was made after reviewing the attrition tables using the two criteria and before any baseline or follow-up analyses were completed.

Study inclusion and exclusion criteria will be finalized during review of the patient attrition table, and prior to any baseline or follow-up analyses.

#### 9.2.4.1 Patient Identification – Eosinophil Subgroup

To be included in the subgroup analysis of patients with at least one eosinophil lab result, patients will be required to meet the patient identification criteria outlined in Section 9.2.4. as well as having at least one eosinophil lab result in the six months prior to the index date (index date -179 days) through 15 days after the index date (index date +15 days). Additionally, the number of patients with  $\ge 1$  eosinophil result in the three months prior the index date (index date -89 days) through to the index date will be identified. The time period for identification of  $\ge 1$  eosinophil result will be determined based on the number of patients identified during these time windows.

Eosinophil test results will be categorized, according to the eosinophil test result closest to the index date during the time period of interest (i.e., with the smallest absolute difference in days between the lab date and the index date), as >300 cells/ $\mu$ L or  $\leq 300$  cells/ $\mu$ L. For multiple eosinophil laboratory results on the same date of service, the highest value will be retained.

c37262534-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 9.2.5 Study visits

Not applicable

**NIS Protocol** 

### 9.2.6 Study discontinuation

Not applicable

#### 9.3 VARIABLES

#### 9.3.1 Exposures

Patients will be assigned to one of the following mutually exclusive study cohorts based on the index pharmacy claim: TIO/OLO or FF/UMEC/VI.

#### 9.3.2 Outcomes

#### 9.3.2.1 Primary outcomes

The following outcomes will be measured in the baseline and follow-up periods. The baseline period will include claims occurring on the index date, except for the index medication claims, which will be included in the follow-up period.

- All-cause health care resource utilization: Indicator variables and counts of physician office visits, hospital outpatient visits, ED visits, "other" (non-inpatient) visits, inpatient stays, and pharmacy claims will be created. Other medical visits are a residual category that includes, but is not limited to, services rendered at independent laboratories, assisted living facilities, and by home health providers. An indicator variable will be created to identify inpatient stays with an acute stay during the inpatient admission. The length of inpatient stays will also be captured. The time to first inpatient stay, the time to first inpatient stay with an acute stay, and the time to first ED visit during follow-up will be captured.
- COPD and/or pneumonia-related health care resource utilization: This utilization will be calculated analogously to all-cause utilization, but restricted to medical claims with a diagnosis for COPD, pneumonia, or acute bronchitis/bronchiolitis in any position (Annex 3) and pharmacy claims for a COPD-related treatment (Annex 3), including COPD-guideline recommended antibiotics (Annex 3).
- **COPD-related health care resource utilization:** This utilization will be calculated analogously to all-cause utilization, but restricted to medical claims with a diagnosis for COPD in any position (Annex 3) and pharmacy claims for a COPD-related treatment (Annex 3), including COPD-guideline recommended antibiotics (Annex 3).

NIS Protocol

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- Pneumonia-related health care resource utilization: This utilization will be calculated analogously to all-cause utilization, but restricted to medical claims with a diagnosis for pneumonia in any position (Annex 3).
- COPD or pneumonia-attributable health care resource utilization: This utilization will be calculated analogously to all-cause utilization, but restricted to medical claims with a diagnosis for COPD, pneumonia, or acute bronchitis/bronchiolitis in the primary position or a diagnosis for acute respiratory failure in the primary position and a diagnosis for COPD, pneumonia, or acute bronchitis/bronchiolitis in a non-primary position (Annex 3) and pharmacy claims for a COPD-related treatment (Annex 3), including COPD-guideline recommended antibiotics (Annex 3).
- All-cause health care costs (insurer + patient paid amounts): Health care costs will be computed from the payer and patient perspective together. This is the actual amount paid to the provider by the health plan plus the patient copay and/or coinsurance amounts, rather than an estimated cost. Total costs will be calculated and presented as the combined pharmacy costs and medical costs. Medical costs will be presented and will include sub-categories of physician office costs, hospital outpatient costs, emergency services costs, inpatient costs, and other costs.
  - Costs will be adjusted to 2020 dollars using the medical care component of the Consumer Price Index (CPI) to reflect inflation between the date of the claim and 2020 [R21-4317]. The final report will include additional columns with the latest available 2021 mid-year CPI adjustment applied to costs for scaling the results as needed.
  - Costs from other payers may be important, particularly for studies involving older patients dually eligible for commercial and Medicare coverage. In consultation with BIPI, this study will NOT incorporate the amounts estimated to be paid by other payers for a total paid or allowable amount [P21-11033].
- COPD and/or pneumonia-related health care costs (insurer + patient paid amounts): These costs will be calculated analogously to the all-cause costs, but restricted to medical claims with a diagnosis for COPD, pneumonia, or acute bronchitis/bronchiolitis in any position (Annex 3) and pharmacy claims for a COPD-related treatment (Annex 3), including COPD-guideline recommended antibiotics (Annex 3).
- COPD-related health care costs (insurer + patient paid amounts): These costs will be calculated analogously to the all-cause costs, but restricted to medical claims with a diagnosis for COPD in any position (Annex 3) and pharmacy claims for a COPD-related treatment (Annex 3), including COPD-guideline recommended antibiotics (Annex 3).

NIS Protocol 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- Pneumonia-related health care costs (insurer + patient paid amounts): These costs will be calculated analogously to the all-cause costs, but restricted to medical claims with a diagnosis for pneumonia in any position (Annex 3).
- COPD or pneumonia-attributable health care costs (insurer + patient paid amounts): These costs will be calculated analogously to the all-cause costs, but restricted to medical claims with a diagnosis for COPD, pneumonia, or acute bronchitis/bronchiolitis in the primary position or a diagnosis for acute respiratory failure in the primary position and a diagnosis for COPD, pneumonia, or acute bronchitis/bronchiolitis in a non-primary position (Annex 3) or pharmacy claims for a COPD-related treatment (Annex 3), including COPD-guideline recommended antibiotics (Annex 3).
- **COPD exacerbations:** Exacerbations will be categorized as moderate or severe and a count of any (severe or moderate), severe, and moderate will be provided. The time to first severe exacerbation, and time to first exacerbation (severe or moderate), during follow-up will be captured. Diagnosis codes that will be used to identify exacerbation-related medical visits are included in <u>Annex 3</u>. COPD-related treatments are listed in <u>Annex 3</u> and COPD-guideline recommended antibiotics are listed in <u>Annex 3</u>. Details of the exacerbation definition are provided in <u>Annex 3</u>.
  - A severe exacerbation will be defined as follows:
  - An inpatient admission or an ER visit with a COPD diagnosis code in the primary position; or
  - An inpatient admission or an ER visit with a diagnosis code for acute respiratory failure in the primary position and a COPD diagnosis code in any position; or
  - An inpatient admission or an ER visit with a diagnosis code for acute respiratory failure in the primary position + an inpatient admission or an ER visit within ±7 days with a COPD diagnosis code in any position.
  - A moderate exacerbation will be defined as follows:
  - An ambulatory (office or outpatient) visit with a COPD diagnosis code in any position + a pharmacy claim for an oral corticosteroid (OCS) prescription within ±7 days of the office/outpatient visit; or
  - An office or outpatient visit with a COPD diagnosis code in any position + a pharmacy claim for COPD-guideline recommended antibiotic prescription within ±7 days of the office/outpatient visit; or
  - An office or outpatient visit with a COPD diagnosis code in any position + a pharmacy claim for an OCS + a pharmacy claim for COPD-guideline recommended antibiotic prescription within ±7 days of the office/outpatient visit.

NIS Protocol 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- Baseline GOLD exacerbation history: Indicator variables will be created to identify patients with no baseline exacerbation or 1 baseline exacerbation not leading to hospitalization (i.e. baseline GOLD A/B) and with ≥2 baseline exacerbations not leading to hospitalization or ≥1 baseline exacerbation leading to hospitalization (i.e. baseline GOLD C/D). These baseline GOLD classification variables will be used to classify the patient population for analysis by exacerbation history.
  - Baseline exacerbation not leading to hospitalization will be defined as follows:
    - An ER visit with a COPD diagnosis code in the primary position; or
    - An ER visit with a diagnosis code for acute respiratory failure in the primary position and a COPD diagnosis code in any position; or
    - An ER visit with a diagnosis code for acute respiratory failure in the primary position + an ER visit within ±7 days with a COPD diagnosis code in any position; or
    - An ambulatory (office or outpatient) visit with a COPD diagnosis code in any position + a pharmacy claim for an oral corticosteroid (OCS) prescription within ±7 days of the office/outpatient visit; or
    - An office or outpatient visit with a COPD diagnosis code in any position + a pharmacy claim for COPD-guideline recommended antibiotic prescription within ±7 days of the office/outpatient visit; or
    - An office or outpatient visit with a COPD diagnosis code in any position + a pharmacy claim for an OCS + a pharmacy claim for COPD-guideline recommended antibiotic prescription within ±7 days of the office/outpatient visit.
  - Baseline exacerbation leading to hospitalization will be defined as follows:
  - An inpatient admission with a COPD diagnosis code in the primary position; or
  - An inpatient admission with a diagnosis code for acute respiratory failure in the primary position and a COPD diagnosis code in any position; or
  - An inpatient admission with a diagnosis code for acute respiratory failure in the primary position + an inpatient admission or an ER visit within ±7 days with a COPD diagnosis code in any position; or
  - An ER visit with a diagnosis code for acute respiratory failure in the primary position + an inpatient admission within ±7 days with a COPD diagnosis code in any position.
- **Pneumonia diagnosis:** Binary indicators will be created to identify patients with a diagnosis of 1) pneumonia or 2) pneumonia or acute bronchitis/bronchiolitis in any position (<u>Annex 3</u>). The time to first pneumonia diagnosis, and time to first pneumonia or acute bronchitis/bronchiolitis diagnosis, during follow-up will also be captured.
- **Pneumonia-related hospitalization:** Binary indicators will be created to identify patients with an acute hospitalization with diagnosis of 1) pneumonia or 2) pneumonia or acute bronchitis/bronchiolitis in any position (Annex 3). The time to first

NIS Protocol Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

pneumonia-related acute hospitalization, and time to first pneumonia- or acute bronchitis/bronchiolitis-related acute hospitalization, during follow-up will also be captured.

• COPD exacerbation and/or pneumonia diagnosis: Binary indicators will be created to identify patients with each of the following composite outcomes: severe COPD exacerbation or an acute hospitalization with a diagnosis of pneumonia in any position, severe COPD exacerbation or an acute hospitalization with a diagnosis of pneumonia or acute bronchitis/bronchiolitis in any position, any COPD exacerbation or pneumonia diagnosis in any position, and any COPD exacerbation or pneumonia diagnosis or acute bronchitis/bronchiolitis diagnosis in any position. Time to event variables will be created for each composite outcome during the follow-up period.

#### 9.3.2.2 Secondary outcomes

**COPD readmission (Centers for Medicare and Medicaid Services [CMS] definition):** COPD readmissions, based on the 2017 CMS specifications as described below [R21-4119], will be captured.

- COPD-related hospitalizations will be identified during the patient's follow-up. Hospitalizations will be classified as COPD-related if they met either of the following 2 criteria:
- ≥1 diagnosis of COPD (Annex 3) in the primary position any time during the acute inpatient stay; or
- ≥1 diagnosis of acute respiratory failure (Annex 3) in the primary position and a diagnosis of acute exacerbation of COPD (Annex 3) in a later position on the same claim during an acute inpatient stay.
- For each qualifying COPD-related hospitalization, an indicator variable will be created to identify if there was a re-admission that started within 30 days of the discharge of the COPD-related hospitalization.
- COPD-related hospitalizations will be required to have at least 30 days of enrollment after the discharge to be included in the analysis, unless readmission and death occur within 30 days of hospital discharge. Hospitalizations that ended within 30 days of the end date will be not included because readmission status cannot be determined accurately.
- COPD-related hospitalizations that ended because the patient discharged themselves against medical advice will be excluded from the analysis, and allcause hospitalizations that included procedures and diagnoses (Annex 3) that are always considered planned (i.e., transplant surgery, maintenance chemotherapy/immunotherapy, and rehabilitation) will not be eligible to be a readmission.



NIS Protocol 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 9.3.3 Covariates

#### 9.3.3.1 Clinical Characteristics

Clinical characteristics will be measured in the baseline period. The baseline period will <u>include</u> claims occurring on the index date, except for the index medication claims, which will be included in the follow-up period.

- Quan-Charlson comorbidity score: A comorbidity score will be calculated based on the presence of diagnosis codes (in any position) on medical claims in the baseline period [R21-4087; R20-2288; R14-4775]. The score is calculated based on a weighted sum of 12 comorbid conditions. The score represents the cumulative likelihood of one-year mortality and serves as a proxy for comorbidity burden. The Quan-Charlson comorbidity score also will be categorized into the following groups: zero, one, two, three, four, and five or more.
  - Charlson Comorbidity Score without COPD: In addition to the standard Charlson comorbidity score, a modified score removing COPD diagnosis codes will be calculated.
- Elixhauser score: The Elixhauser score will be calculated based on the presence of diagnosis codes (any position) on medical claims during the baseline period [R13-3591]. Elixhauser comorbidities will be consolidated into a single numeric score to summarize disease burden [R21-4090] The score is calculated based on a weighted sum of 31 comorbid conditions. The score represents the likelihood of hospital mortality, and serves as a proxy for comorbidity burden, similar to the Charlson score.
  - Elixhauser score without COPD: A modified score removing COPD diagnosis codes will also be calculated.
- **COPD Severity Score:** The COPD Severity score will be calculated as a weighted sum of the individual components listed in <u>Table 1</u> during the baseline period [<u>R21-4086</u>]. The COPD Severity score is a validated measure of COPD severity based on treatments.

NIS Protocol

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### Table 1 COPD Severity Score Components

| Component (input from claims) | How Identified in Claims |
|---|---|
| Count of exacerbations | See definition for COPD Exacerbations above |
| Oxygen therapy – current | CPT, HCPCS, ICD-10, ICD-9 and revenue codes |
| Length of stay for COPD-<br>attributable inpatient<br>visits | ICD-9 or ICD-10 code for COPD in the primary position or a code for acute respiratory failure in the primary position and a code for COPD in a non-primary position |
| Emphysema | ICD-9 or ICD-10 code in any position on a medical claim |
| Spirometry testing | See Spirometry Testing, below |
| Pulmonologist visits | Physician specialty |
| Use of SAMAs (including SABA/SAMA combination) | See Medication Utilization, above |
| Use of oral corticosteroids | See Medication Utilization, above |
| Use of inhaled corticosteroids | See Medication Utilization, above |
| Use of SABAs (including SABA/SAMA combination) | See Medication Utilization, above |
| Use of long-acting bronchodilators | See Medication Utilization, above |
| Mean age | Age as of baseline year |

- Additional comorbid conditions: Additional comorbid conditions, including allergic rhinitis, anxiety (narrow and broad), arrhythmia, atrial fibrillation (narrow and broad), acute sinusitis, candidiasis, cataracts, chronic sinusitis, chronic rhinitis, congestive heart failure, depression, diabetes (type I and II), dyspnea, hypertension, ischemic heart disease, metabolic syndrome (including individual components), myocardial infarction, osteoporosis, pulmonary fibrosis, peripheral vascular disease, peptic ulcer/GERD, renal disease, sleep apnea, stroke, pneumonia, and pneumonia or acute bronchitis/bronchiolitis will also be identified based on the presence of a diagnosis code in any position on a medical claim (Annex 3).
- Oxygen therapy: Evidence of oxygen use will be captured in the baseline period based on diagnosis (ICD-9, ICD-10), procedure (HCPCS, CPT, ICD-9) and revenue codes for oxygen therapy (Annex 3).

Stiolto vs Trelegy V1.0 04 May

021

NIS Protocol

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- Baseline respiratory medication utilization: Indicator variables for respiratory medication classes and selected individual respiratory medications will be based on both pharmacy and medical claims (nebulizer treatments may appear in medical claims). Medication classes will include: LAMAs (alone; overall and separately), LABAs (alone), ICS (alone), ICS/LABA single inhaler combination medications, SAMAs (alone), SABAs (alone), SAMA/SABA single inhaler combination medications, any rescue (SAMA alone, SABA alone, or SAMA/SABA single inhaler combination medications), methylxanthines, phosphodiesterase-4 (PDE-4) inhibitors and oral corticosteroids (OCS). Baseline medication use variables will exclude claims which make up the index therapy assignment. Number of fills by class will also be captured. Indicator variables will be created to identify patients who are naïve to long-acting bronchodilators (free or fixed dose LAMAs or LABAs) and to long-acting bronchodilators plus inhaled corticosteroids (free or fixed dose LAMAs, LABAs, and ICSs) at index.
- Index provider specialty: The specialty of the provider on the index prescription fill will be captured. If no provider specialty is recorded on the index prescription fill, the provider specialty from the most recent COPD-related visit on or prior to the index date will be captured. An indicator variable will identify if the provider specialty was determined from the index pharmacy claim. Provider specialty will be classified as one of the following: pulmonology, primary care [family practice, general practice, and geriatrics], internal medicine, allied health professional, cardiology, other specialty, and unknown specialty. If claims for more than one provider occur on the date used to classify the provider's specialty, the hierarchy of categories listed above will be used to pick a single provider specialty.
- Pulmonology visit within 30 days of index date: An indicator variable will be created to identify patients with a pulmonologist visit within 30 days prior to and excluding the index date.
- **Spirometry testing:** Indicator and count variables will be created to identify patients with lung function testing (<u>Annex 3</u>). A count of spirometry tests during the baseline period will be created.
- Early adopter of index medication: An indicator variable will be created to identify patients with an index date within 90 days of FDA approval of the medication. The FDA approval date is specific to the index therapy: Stiolto Respimat (TIO/OLO) was FDA approved on 21 May 2015 and Trelegy Ellipta (FF/UMEC/VI) was FDA approved on 18 September 2017.
- Evidence of tobacco use: An indicator variable will be created to identify patients with evidence of current or prior tobacco use based on diagnosis codes (Annex 3) or pharmacy fills for smoking cessation treatments (bupropion, varenicline tartrate, or nicotine inhalation system).

c37262534-01 

NIS Protocol

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 9.3.3.2 Patient Characteristics

Patient characteristics will be measured as of the index date, or the first available claim after the index date with valid values for each of the characteristics. Approval through the data disclosure analysis process is required for inclusion of socioeconomic data (i.e., race/ethnicity) and resource scare areas. Approval is not guaranteed. It may be necessary to modify or remove some variables or analytic table templates in order to preclude identification of individual patients and protect proprietary health plan information.

- Index year: The year of the patient's index date will be identified.
- Seasonality: The month of the patient's index date will be identified and classified as fall (September, October, November), winter (December, January, February), spring (March, April, May), or summer (June, July, August).
- Age: Age will be defined as of the index year
- **Age groups:** Patients will be assigned to one of the following age groups: 40-49, 50-59, 60-64, 65-69, 70-74 and 75+
- **Gender:** Gender will be captured from enrollment data; patients with undefined gender will be removed from the study sample
- Race/ethnicity: Race/ethnicity information will be captured from the linked consumer sociodemographic data and categorized as follows: White, African-American/Black, Asian, Hispanic, or unknown (unknown includes missing). This variable depends on the availability of data within the sociodemographic data and will be missing for some patients.
- **Insurance type:** Whether the patient was covered under a commercial or Medicare Advantage health plan will be captured
- Plan type: Plan type will be categorized as Exclusive Provider Organization (EPO), Health Maintenance Organization (HMO), Point of Service (POS), Preferred Provider Organization (PPO), Individual and Other
- **Geographic region:** The US region in which the study patient is enrolled in a health plan will be determined and reported and states will be categorized into five geographic regions in accordance with the US Census Bureau's region designations; the five health plan regions are presented in the table below. Patients categorized into "other" will be excluded from the study.
- **Resource scarce area:** Health professional shortage areas (HPSAs) will be identified based on the Health Resources and Services Administration designation of geographic regions with a shortage of providers to meet the needs of the population [R21-4295].

NIS Protocol Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 2 Health Plan Regions

| Region | State |
|---|---|
| Northeast | CT, MA, ME, NH, RI, VT, NJ, NY, PA |
| Midwest | IL, IN, MI, OH, WI, IA, KS, MN, MO, ND, NE, SD |
| South | DC, DE, FL, GA, MD, NC, SC, VA, WV, AL, KY, MS, TN, AR, LA, OK, TX |
| West | AZ, CO, ID, MT, NM, NV, UT, WY, AK, CA, HI, OR, WA |

#### 9.4 DATA SOURCES

when combined with Medicare Part D coverage.



In 2018, the D included claims for approximately 19% of the US commercially enrolled population and approximately 21% of the Medicare Advantage population (commonly referred to as the Medicare Advantage program [Medicare Part C]) through an offering associated with Medicare Advantage enrollees choose to receive all of their health care services through a provider organization in lieu of Medicare Part A/B coverage (commonly referred to as Medicare Fee for Service). These plans are referred to as MAPD

Underlying information is geographically diverse across the United States and enrollees are fairly representative of the US population. Because the D is a closed system, patients retain a single identifier within the system and can be tracked as they change plans, or as they disenroll and reenroll over time.

Claims for pharmacy services are typically submitted electronically by the pharmacy at the time prescriptions are filled. The claims history is a profile of all outpatient prescription pharmacy services provided and covered by the health plan. Pharmacy claims data include drug name, dosage form, drug strength, fill date, days of supply, financial information, and de-identified patient and prescriber codes, allowing for longitudinal tracking of medication refill patterns and changes in medications. Pharmacy claims are typically added to the research database within six weeks of dispensing.

Medical claims or encounter data are collected from all available health care sites (inpatient hospital, outpatient hospital, emergency department, physician's office, surgery center, etc.) for virtually all types of provided services, including specialty, preventive and office-based treatments. Medical claims and coding conform to insurance industry standards. Claims for ambulatory services submitted by individual providers, such as physicians, use the Health

c37262534-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Care Financing Administration (HCFA)-1500 or Centers for Medicare and Medicaid Services (CMS)-1500 formats. Claims for facility services submitted by institutions, e.g., hospitals, use the Uniform Billing (UB)-82, UB-92, UB-04, or CMS-1450 formats. Medical claims include: multiple diagnosis codes recorded with the International Classification of Diseases, Ninth Revision, Clinical Modification (ICD-9-CM) and International Classification of Diseases, Tenth Revision, Clinical Modification (ICD-10-CM) diagnosis codes; procedures recorded with ICD-9-CM and ICD-10-CM procedure codes, Current Procedural Terminology (CPT), or Health care Common Procedure Coding System (HCPCS) codes; site of service codes; provider specialty codes; revenue codes (for facilities); paid amounts; and other information. Typically, facility claims do not include medications dispensed in hospital. Approximately six months following the delivery of services is required for complete medical data.

#### 9.4.2 Laboratory Results

**NIS Protocol** 

Outpatient laboratory test results are available for subpopulations of the research database. Standard LOINC coding is used to define specific tests and results. Test results data can be linked to the other health care utilization and pharmacy claims data in the research database. Results included in the database are typically from blood-based tests (e.g., LDL, HbA1c) that are sent for processing to one of several laboratory facilities in the country that provide services to enrollees in the health plan. For common blood-based tests such as lipids and HbA1c, results are typically available for approximately 40-50% of tests performed. However, this proportion varies by test and by disease state. In addition, study requirements such as the timing of the laboratory result or the requirement of multiple results to assess change over time will be available for smaller subsets of the study population. Results dating back to 2000 are available for research.

Laboratory results are typically added to the research database within three to six months of administration of the test.

#### 9.5 STUDY SIZE

Using claims data for commercial and Medicare Advantage health plan enrollees we identified 5,717 and 17,733 patients who initiated treatment with TIO/OLO or FF/UMEC/VI, respectively, between 01 January 2018 and 31 July 2019. These patients had 12-months of baseline and ≥30 days of follow-up continuous enrollment with both medical and pharmacy coverage. This count is for informational purposes only and may not represent the actual number of patients to be utilized in the study. Application of other inclusion and exclusion criteria required for this study or other factors may reduce the sample size.

#### 9.6 DATA MANAGEMENT

Not applicable

Stiolto vs Trelegy V1.0 04 May

2021

NIS Protocol 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 9.7 DATA ANALYSIS

All statistical analyses will be performed by using using , ) or later. The conventional significance level  $\alpha$ =0.05 will be used to determine statistical significance.

#### 9.7.1 Comparison of TIO/OLO Initiators

Given the difference in FDA approval dates (May 2015 for TIO/OLO and September 2017 for FF/UMEC/VI) and concerns about retaining adequate sample size for the analyses the following stepwise approach will be implemented to finalize the patient identification period

- 1) In the overall population, TIO/OLO initiators from May 2015 December 2017 will be compared to TIO/OLO initiators from January 2018 November 2019 on a prespecified list of characteristics including:
  - Demographics (age in years, gender, geographic region, insurance type [commercial vs. MAPD], prescriber specialty, pulmonologist visit within 30 days prior to and excluding the index date)
  - Clinical comorbidities (diabetes, hypertension, ischemic heart disease, Elixhauser score without COPD)
  - COPD severity proxies (dyspnea, oxygen therapy, maintenance naïve, no baseline exacerbation or 1 baseline exacerbation not leading to hospitalization, ≥2 baseline exacerbations not leading to hospitalization or ≥1 baseline exacerbation leading to hospitalization)
- 2) If TIO/OLO initiators from before and after FF/UMEC/VI approval are well balanced (i.e., standardized difference ≤10%) across all characteristics outlined in step one, the start of the patient identification period will remain 01 June 2015.
- 3) If TIO/OLO initiators from before and after FF/UMEC/VI approval have standardized differences >10% on one to three characteristics listed in step one, those characteristics will be included as covariates in post-match multivariable regression analysis.
- 4) If TIO/OLO initiators from before and after FF/UMEC/VI approval have standardized differences >10% on four or more characteristics listed in step one, the start of the patient identification period will be moved from 01 June 2015 to 01 January 2018.

#### 9.7.2 Main analysis

Not applicable

c37262534-01  **NIS Protocol** 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 9.7.3 **Primary Objectives**

## 9.7.3.1 Descriptive Analysis

Baseline categorical variables will be presented as numbers and percentages and baseline continuous variables will be presented as means, standard deviations, medians, and interquartile ranges. Follow-up variables will be presented as population annualized averages to account for the variable follow-up duration (minimum 1 month, maximum 12 months). Population annualized averages will be calculated as ([sum of all utilization or cost for all individuals during the follow-up period]/[sum of all follow-up time in days for all individuals])\*365. Wald 95% confidence intervals (CI) will be provided for annualized population averages using the Taylor expansion to estimate the standard error. The numerator and denominator of the population annualized average equation and the 95% CI will be presented. Per patient per month calculations will not be performed. Appropriate statistical tests comparing treatment cohorts (e.g., t-test, chi-square test) will be used based on the distribution of the measure (Table 3)

Bivariate comparisons of patient demographics and baseline characteristics will be provided for the TIO/OLO and FF/UMEC/VI cohorts prior to PSM. Following the matching procedure, bivariate comparisons of demographics and baseline characteristics will be provided to assess the success of the matching procedure, and comparisons of outcomes will be provided to assess the impact of initiating treatment with TIO/OLO vs FF/UMEC/VI. Appropriate tests comparing the TIO/OLO cohort and the FF/UMEC/VI cohort (e.g., standardized differences, McNemar's tests, paired t-tests, sign tests) (Table 3) will be used based on the distribution of the measure. Patients not matched will be excluded from the postmatch analysis. In addition to presenting the results stratified by treatment cohort (TIO/OLO vs. FF/UMEC/VI), the results will be presented stratified by treatment cohort among the following populations: maintenance naïve (patients with no baseline maintenance medication [no free or fixed dose LAMA, LABA, or ICS]); no exacerbation (patients with no baseline exacerbation); no exacerbation or one exacerbation not leading to hospitalization (i.e., baseline GOLD A/B); at least two exacerbations not leading to hospitalization or at least one exacerbation leading to hospitalization [i.e., baseline GOLD C/D]). Results also will be presented for the subset of the population with at least one eosinophil laboratory result.

001-

NIS Protocol Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 3 Statistical Testing by Descriptive Variable Type

| Variable type | Baseline | Variable follow-up comparisons between study cohorts |
|---|---|---|
| Categorical | Pearson's chi-square<br>Fisher's exact test | Kaplan-Meier |
| Continuous | Independent samples t-test<br>Wilcoxon-Mann Whitney<br>test | Population annualized averages |
| Time-to-event variables | N/A | Incidence rate or Kaplan-Meier |

#### 9.7.3.2 Kaplan Meier Analysis

Kaplan–Meier (KM) analysis will be used to estimate time to first COPD exacerbation (any, severe), time to first pneumonia diagnosis, and time to first pneumonia hospitalization. When KM analysis is conducted, results will include censored-adjusted percentage of patients who have had at least one event of interest (i.e., COPD exacerbation, pneumonia diagnosis, pneumonia hospitalization) at pre-specified time periods of interest (e.g., 1 month, 3 months, 6 months). In addition, the median (and 25th and 75th percentile) time to event and the 95% confidence interval around the median (and 25th and 75th percentile) will be reported. A p-value will be calculated using the log rank test to examine if the distribution of outcomes among patients in the TIO/OLO cohort versus the FF/UMEC/VI cohort are different. In addition to presenting results for the overall TIO/OLO versus FF/UMEC/VI comparison, KM analysis also will be conducted among the following populations: maintenance naïve; no exacerbation; no exacerbation or one exacerbation not leading to hospitalization; at least two exacerbations not leading to hospitalization with at least one exacerbation leading to hospitalization; subset of the population with at least one eosinophil laboratory result.

#### 9.7.3.3 Number Needed to Treat

Based on the descriptive analysis results, the number of FF/UMEC/VI patients that would instead need to be treated (i.e., number needed to treat [NNT]) with TIO/OLO to avoid one event (e.g., exacerbation of COPD) will be calculated for key outcomes. The NNT will be calculated using the following equation: 1/(Event RateFF/UMEC/VI – Event RateTIO/OLO). Rates will be derived from the annualized Kaplan-Meier analyses.

#### 9.7.3.4 Multivariable Analysis (Optional)

Multivariable regression will be included in the analysis if either TIO/OLO initiators from before and after FF/UMEC/VI approval have standardized differences of >10% on one to three characteristics listed in <u>Section 9.7.1</u>. or if there are standardized differences of >10%

c37262534-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

between the TIO/OLO and FF/UMEC/VI cohorts after PSM. If multivariable model is included, the appropriate regression model will be selected based on the distribution of the measure. Because health care costs are often skewed, cost measures may be modeled using Manning and Mullahy's formulation. This method avoids potential difficulties introduced by transformation and retransformation of the dependent variable. Specifically, the outcome is modeled employing a GLM with a gamma distribution and log link. Exponentiated coefficients from a GLM are estimated cost ratios. Cost ratios, 95% confidence intervals, and p-values will be presented for each covariate included in the final model. For ease of interpretation and comparison with the bivariate results, the average cost will be predicted for each cohort using recycled predictions. Cox proportional hazard modeling may be used for the exacerbation and pneumonia outcomes.

## 9.7.4 Secondary Objective

NIS Protocol

#### 9.7.4.1 COPD Readmission CMS Definition

• CMS-based readmission analysis will not be conducted for the subgroup analysis among patients with available eosinophil lab results.

A hospitalization-level analysis will be performed to examine how many COPD-related hospitalizations resulted in an all-cause inpatient readmission within 30 days of discharge. The sample size for this analysis will be the number of qualifying COPD-related hospitalizations that occur during the follow-up, and consequently a patient may contribute 0, one, or more than one observation to the analysis. A patient with no COPD-related hospitalizations will not contribute any observations to the analysis, and a patient with two COPD-related hospitalizations five months apart may contribute two observations to the analysis. The number and percent of follow-up COPD-hospitalizations that result in an allcause readmission will be calculated. An unmatched descriptive analysis will be conducted because the unit of analysis will be hospitalizations, not patients. Logistic regression will be conducted to determine if the adjusted odds of a readmission are different for hospitalizations among TIO/OLO initiators versus hospitalizations among FF/UMEC/VI initiators. The logistic regression model will include the propensity score model covariates, plus an additional baseline readmission covariate. A variable will be created to identify if the person associated with the hospitalization had: 1) at least one baseline COPD hospitalization that resulted in a readmission; 2) at least one baseline COPD hospitalization but none of them resulted in a readmission; 3) no baseline COPD-related hospitalization. The logistic regression model will account for clustering since patients could contribute multiple observations (i.e., multiple qualifying COPD hospitalizations).



**NIS Protocol** 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 9.8 LIMITATIONS OF THE RESEARCH METHODS

An inherent limitation of observational studies involving non-random allocation of treatment is a form of selection bias called 'confounding by indication'. With this type of selection bias, the underlying patient characteristics associated with a certain treatment (i.e., TIO/OLO or the comparator) may influence the outcome under study. The current study proposes to address the bias from confounding by indication with PSM. The aim of PSM is to balance two non-equivalent groups on observed baseline characteristics to be able to obtain less biased estimates of treatment effects. This balancing can be achieved by either matching study patients in comparison groups on propensity scores, weighting for propensity scores, or adjusting for propensity scores in the analysis. This therefore ensures that the distribution of characteristics is the same for patients who initiate TIO/OLO and FF/UMEC/VI.

Second, an "on-treatment" analysis is planned in which patients will be censored at the time of discontinuation of the index medications or initiation of another COPD maintenance medication (as well as for disenrollment from the health plan, 12-months following the index date, or the end of the study period). Therefore, the conclusions from this study will be applicable to patients who initiate and remain on the study treatments, rather than the broader population of patients who initiate one of the study treatments (i.e., an intention to treat analysis) and therefore is potentially prone to survival bias. By censoring at the time of discontinuation of the index medication rather than the discontinuation date + 30 days outcomes that occur right after medication discontinuation, which may be related to the index medication, are not captured.

Third, patients with one or more days of free or fixed dose LAMA/LABA maintenance therapy in the six month pre-index period will be excluded from the study sample. The GOLD 2018 and 2019 recommendations maintain that TT should only be used as an escalation step following treatment with LAMA and LABA or LABA and ICS. Thus, patients initiating FF/UMEC/VI in this study, will be a subset of TT initiators who are not following the GOLD recommendations.

Fourth, the patient identification period starts at the FDA approval of TIO/OLO (May 2015) rather than the FDA approval of FF/UMEC/VI (September 2017). By design, patient index year will not be included/ as a matching variable for the PSM models because there will be no FF/UMEC/VI initiators to match in the first part of the patient identification period. TIO/OLO initiators from May 2015 – December 2017 will be compared to TIO/OLO initiators from January 2018 – November 2019 on a prespecified list of characteristics as outlined in Section 9.7.1. If there are differences between TIO/OLO initiators from before and after FF/UMEC/VI approval the start of the patient identification period will be moved to 01 January 2018. Index year may be included in multivariable regression analysis to determine if the index year (i.e., initiation date) is a confounder of the association between treatment and outcomes. If index year is a significant predictor in the multivariable regression model, sample selection may be restricted to patients with an index date following FF/UMEC/VI launch or the sample may be restricted to a time period where index year is not a significant covariate in the multivariable regression model.
c37262534-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Finally, claims data are subject to certain limitations. In addition to miscoding, omissions and/or rule-out diagnoses, the presence of a claim for a filled prescription does not indicate that the medication was consumed or that it was taken as prescribed, and any medications filled over-the-counter or provided as samples by the physician will not be observed in the claims data. It also lacks some lifestyle behaviors and clinically relevant characteristics including lung function, smoking status/history, symptom burden that may impact disease progression and in turn the outcome metrics. Data on physician decision-making process on treatment choices is also unavailable and may impact our comparison of an initial vs. a next-in-line treatment. Relying on pharmacy claims for switch and discontinuation definitions will miss patients who use nebulized medications captured via medical claims and may preemptively censor adherent patients. Finally, as with all claims-based analyses, study results may not be generalizable to those with non-commercial or MAPD health insurance.

#### 9.9 OTHER ASPECTS

None

**NIS Protocol** 

### 9.9.1 Data quality assurance

A quality assurance audit/inspection of this study may be conducted by the sponsor or sponsor's designees or by Institutional Review Board (IRBs) / Independent Ethics Committee (IECs) or by regulatory authorities. The quality assurance auditor will have access to all medical records, the investigator's study-related files and correspondence, and the informed consent documentation of this study.

### 9.9.2 Study records

9.9.2.1 Source documents

Not applicable

NIS Protocol 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 10. PROTECTION OF HUMAN SUBJECTS

The study will be carried out in compliance with the protocol, the principles laid down in the Declaration of Helsinki, Guidelines for Good Pharmacoepidemiology Practice (GPP), and the relevant BI Standard Operating Procedures (SOPs). Standard medical care (prophylactic, diagnostic and therapeutic procedures) remains the responsibility of the treating physician of the patient.

# 10.1 STUDY APPROVAL, PATIENT INFORMATION, AND INFORMED CONSENT

This NIS will be initiated only after all required legal documentation has been reviewed and approved by the respective Institutional Review Board (IRB)/Independent Ethics Committee (IEC) and Competent Authority (CA) according to national and international regulations. The same applies for the implementation of changes introduced by amendments.

Prior to patient participation in the study, written informed consent must be obtained from each patient (or the patient's legally accepted representative) per GPP and according to the regulatory and legal requirements of the participating country, if applicable.

### 10.2 STATEMENT OF CONFIDENTIALITY

No patient's identity or medical records will be disclosed for the purposes of this study except in compliance with applicable law.

NIS Protocol 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 11. MANAGEMENT AND REPORTING OF ADVERSE EVENTS/ADVERSE REACTIONS

# 11.1 ADVERSE EVENT AND SERIOUS ADVERSE EVENT COLLECTION AND REPORTING

## Collection of AEs

Not applicable based on secondary use of data without any potential that any employee of BI or agent working on behalf of BI will access individually identifiable patient data.

Stiolto vs Trelegy V1.0 04 May

2021

**NIS Protocol** 

c37262534-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 12. PLANS FOR DISSEMINATING AND COMMUNICATING STUDY RESULTS

The rights of the investigator and of the sponsor with regard to publication of the results of this study are described in the investigator contract. As a general rule, no study results should be published prior to finalization of the Study Report.

Stiolto vs Trelegy V1.0 04 May

2021

13. REFERENCES

## 13.1 PUBLISHED REFERENCES

- P20-06571 Palli SR, Frazer M, DuCharme M, Buikema AR, Anderson AJ, Franchino-Elder J. Differences in Real-World Health and Economic Outcomes Among Patients with COPD Treated with Combination Tiotropium/Olodaterol Versus Triple Therapy. J Manag Care Spec Pharm. 2020;26(10):1363-1374.
- R18-1532 Lipson DA, Barnhart F, Brealey N, et al. Once-Daily Single-Inhaler Triple versus Dual Therapy in Patients with COPD. N Engl J Med. 2018;378(18):1671-1680.
- R21-4089 Lipson DA, Crim C, Criner GJ, et al. Reduction in All-Cause Mortality with Fluticasone Furoate/Umeclidinium/Vilanterol in Patients with Chronic Obstructive Pulmonary Disease. Am J Respir Crit Care Med. 2020;201(12):1508-1516.
- R21-4088 Bogart MR, Hopson SD, Shih HC, Stanford RH, Coutinho AD. COPD exacerbation costs in the IMPACT study: a within-trial analysis. Am J Manag Care. 2020;26(5):e150-e154.
- R12-1912 Rosenbaum PR, Rubin DB. The central role of the propensity score in observational studies for casual effects. Biometrika. 1983;70(1):41-55.
- R21-4317 U.S. Department of Labor BoLS. Consumer Price Index. Medical Care. Series ID: CUUR0000SAM. http://data.bls.gov/cgi-bin/surveymost?cu.
- P21-11033 Frytak JR, Henk HJ, Zhao Y, Bowman L, Flynn JA, Nelson M. Health service utilization among Alzheimer's disease patients: evidence from managed care. Alzheimers Dement. 2008;4(5):361-367.
- R21-4119 2017 Condition-Specific Measures Updates and Specifications Report Hospital-Level 30-Day Risk-Standardized Readmission Measures. Yale New Haven Health Services Corporation/Center for Outcomes Research & Evaluation (YNHHSC/CORE).
- R21-4087 Bayliss EA, Ellis JL, Shoup JA, Zeng C, McQuillan DB, Steiner JF. Association of patient-centered outcomes with patient-reported and ICD-9-based morbidity measures. Ann Fam Med. 2012;10(2):126-133.
- R20-2288 Quan H, Li B, Couris CM, et al. Updating and validating the Charlson comorbidity index and score for risk adjustment in hospital discharge abstracts using data from 6 countries. Am J Epidemiol. 2011;173(6):676-682.
- R14-4775 Quan H, Sundararajan V, Halfon P, et al. Coding algorithms for defining comorbidities in ICD-9-CM and ICD-10 administrative data. Med Care. 2005;43(11):1130-1139.

c37262534-01 

**NIS Protocol** 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

R13-3591 Elixhauser A, Steiner C, Harris DR, Coffey RM. Comorbidity measures for use with administrative data. Med Care. 1998;36(1):8-27.

R21-4090 van Walraven C, Austin PC, Jennings A, Quan H, Forster AJ. A modification of the Elixhauser comorbidity measures into a point system for hospital death using administrative data. Med Care. 2009;47(6):626-633.

R21-4086 Wu EQ, Birnbaum HG, Cifaldi M, Kang Y, Mallet D, Colice G. Development of a COPD severity score. Curr Med Res Opin. 2006;22(9):1679-1687.

R21-4295 Health Resources & Services Administration. Data Downloads. Shortage Areas. https://data.hrsa.gov/data/download. Accessed February 02, 2021.

c37262534-01 

**NIS Protocol** Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## ANNEX 1. LIST OF STAND-ALONE DOCUMENTS

None

Stiolto vs Trelegy V1.0 04 May 2021 MCS-90-118\_RD-23 (1.0) / Saved on: 25 Nov 2019

c37262534-01 

**NIS Protocol** Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## ANNEX 2. ENCEPP CHECKLIST FOR STUDY PROTOCOLS

NA

Stiolto vs Trelegy V1.0 04 May 2021 MCS-90-118\_RD-23 (1.0) / Saved on: 25 Nov 2019

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## **ANNEX 3. ADDITIONAL INFORMATION**

Table 1. COPD-related Respiratory Medications and Classes

| Drug Class | Subclass | Medication |
|---|---|---|
| Maintenance | | aclidinium |
| medications | Inhaled long-acting anti- | glycopyrrolate |
| | muscarinic | revefenacin |
| | agents (LAMA) | tiotropium |
| | | umeclidinium |
| | | arformoterol |
| | | formoterol |
| | Long-acting β-agonists (LABA) | indacaterol |
| | | olodaterol |
| | | salmeterol |
| | | beclomethasone |
| | | budesonide (both inhaler and nebulizer) |
| | | ciclensonide |
| | Inhaled corticosteroids (ICS) | flunisolide |
| | | fluticasone |
| | | mometasone |
| | | triamcinolone |
| | | aclidinium/formoterol |
| | | glycopyrrolate/formoterol |
| | Inhaled LAMA/LABA combination | indacaterol/glycopyrrolate |
| | Comomuton | tiotropium/olodaterol |
| | | umeclidinium/vilanterol |
| | | budesonide/formoterol |
| | Inhaled ICS/LABA | fluticasone/salmeterol |
| | combination | fluticasone/vilanterol |
| | | mometasone/formoterol |
| | Inhaled ICS/LABA/LAMA | Budesonide/glycopyrrolate/formoterol |

001-

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Drug Class | Subclass | Medication |
|---|---|---|
| | combination | fumarate <sup>1</sup> |
| | | Fluticasone/umeclidinium/vilanterol |
| | | aminophylline |
| | Methylxanthines (intravenous, oral) | dyphylline |
| | (martinous, orar) | theophylline |
| | PDE-4 inhibitor (oral) | roflumilast |
| Rescue | | albuterol |
| medications | | bitolterol |
| | | isoetharine |
| | Short-acting β-agonists (SABA) (inhalation, oral) | isoproterenol |
| | (SADA) (Illialation, oral) | levalbuterol |
| | | metaproterenol |
| | | pirbuterol |
| | Short-acting anti-muscarinic Agents (SAMA) (inhalation) | ipratropium |
| | SAMA/SABA (inhalation) | ipratropium/albuterol |
| | | betamethasone |
| | | dexamethasone |
| | 0-1 | hydrocortisone |
| | Oral corticosteroids (OCS) <sup>2</sup> | methylprednisolone |
| | | prednisolone |
| | | prednisone |

1This medication was FDA approved for maintenance treatment of COPD on 24 July 2020, which is outside of the study time period, and will not be included in this study.

2Including tablets, oral solutions, alivirs, etc. Injectable corticosteroid medications will not

2Including tablets, oral solutions, elixirs, etc. Injectable corticosteroid medications will not be included.

001-

**NIS Protocol** Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### **COPD Guideline-recommend Antibiotic Medications**

| <b>Drug Category</b> | Drug Class | Medication |
|---|---|---|
| COPD Guideline- | | cefaclor |
| recommended Antibiotics <sup>1</sup> | | cefdinir |
| | | cefditoren |
| | | cefepime |
| | Cephalosporins | cefpodoxime |
| | | cefprozil |
| | | ceftibuten |
| | | ceftriaxone |
| | | cefuroxime |
| | Macrolides | azithromycin |
| | Wacrondes | clarithromycin |
| | | amoxicillin |
| | Penicillins | amoxicillin/potassium |
| | | piperacillin/tazobactam |
| | Quinolones | levofloxacin |
| | | moxifloxacin |
| | Sulfonamide combinations | sulfamethoxazole/trimethoprim |
| | Tetracyclines | doxycycline |

<sup>1</sup>The American Thoracic Society (2017) and Global Initiative for Chronic Obstructive Lung Disease (2020) guidelines recommend that antibiotics for acute exacerbation of chronic bronchitis be selected based on local sensitivity patterns. For more specific recommendations, The Sanford Guide to Antimicrobial Therapy (2020) was referenced.

#### **COPD Exacerbation Definition**

- **Exacerbation Hierarchy:** Exacerbation events will be classified as severe or moderate according to the highest severity contributing event.
- Exacerbation Episodes: Exacerbations occurring within 14 days of each other will be considered a single exacerbation episode and will be classified according to the highest severity contributing event.
- Episode Length: The start date of the exacerbation episode will be the service date of the first event (medical encounter or pharmacy fill for an OCS or antibiotic). The end date of the exacerbation episode will be defined as the last observed exacerbation event date (or discharge date if an inpatient event) + 14 days.

c37262534-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## **Single Event Episode**

**NIS Protocol** 

• In a single event episode, the exacerbation begins with the earliest occurrence of these events: COPD exacerbation defined inpatient admission, ER visit, ambulatory visit, or corticosteroid or antibiotic dispensing as defined in <a href="Section 9.3.2.1">Section 9.3.2.1</a>. In a single event episode, the exacerbation ends 14 days from the start of the event, hospital discharge, or following the OCS or antibiotic dispensing, whichever is later.

**Episode Start date** = service date of a qualifying event (inpatient admission, ED visit, ambulatory visit, or OCS or antibiotic dispensing).

- If the qualifying event is a hospitalization, the start date is the admission date.
- If the qualifying event is an ED visit, the start date is the service date.
- If the qualifying event is an ambulatory visit or an OCS or antibiotic dispensing, the start date is the earliest of the associated medical visit or medication dispensing date.

## **Episode End Date**

- If the qualifying event is a hospitalization: discharge date + 14 days
- If the qualifying event is an ER visit: start date + 14 days
- If the qualifying event is an ambulatory visit or an OCS or antibiotic dispensing: the latest of the medical visit or medication dispensing + 14 days
- If the Episode End Date is after the end of follow-up, then set an additional flag **CENSORED**=1.
- NOTE: Under this definition, it is possible for the runout of a medication to exceed the End Date.

#### MULTIPLE EVENT EPISODES

If another qualifying event occurs before the episode End Date, then the episode is extended. The date of the second event is used to reset the End Date per the definition above, using information from this second event. The process continues until a 14-day period with no exacerbation qualifying events occur. The End Date is set (as defined above).

• **Episode Length**: (End date – Start date) + 1


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


Stiolto vs Trelegy V1.0 04 May 2021 MCS-90-118\_RD-23 (1.0) / Saved on: 25 Nov 2019 001-

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


Stiolto vs Trelegy V1.0 04 May 2021 MCS-90-118\_RD-23 (1.0) / Saved on: 25 Nov 2019 001-


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


Stiolto vs Trelegy V1.0 04 May 2021 MCS-90-118\_RD-23 (1.0) / Saved on: 25 Nov 2019 001-

001-

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


Stiolto vs Trelegy V1.0 04 May 2021 MCS-90-118\_RD-23 (1.0) / Saved on: 25 Nov 2019


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


Stiolto vs Trelegy V1.0 04 May 2021 MCS-90-118\_RD-23 (1.0) / Saved on: 25 Nov 2019 001-


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


Stiolto vs Trelegy V1.0 04 May 2021 MCS-90-118\_RD-23 (1.0) / Saved on: 25 Nov 2019 001-


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


Stiolto vs Trelegy V1.0 04 May 2021 MCS-90-118\_RD-23 (1.0) / Saved on: 25 Nov 2019

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


001-

| of implanted |
|----------------|
| or implanted |
| ment of CSF |
| opacemaker |
| ed nervous |
| f right breast |
| f left breast |
| f unsp breast |
| catheter |
| f oth devices |
| funspecified |
| ph Vein, |
| oh Vein, Open |
| Iarrow into |
| eriph Vein, |
| eriph Vein, |
| Periph Vein, |
| Periph Vein, |
| lood Stem |


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


001-

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


001-

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


001-

**NIS Protocol** 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


**NIS Protocol** 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


**NIS Protocol** 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


**NIS Protocol** 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


**NIS Protocol** 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


001-


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


**NIS Protocol** 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


**NIS Protocol** 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


**NIS Protocol** 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


001-

**NIS Protocol** 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


001-

**NIS Protocol** 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


001-

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


001-

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


001-

**NIS Protocol** 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


001-

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


| ICD-10 Drug or chemical induced diabetes mellitus with diabetic peripheral angiopathy with gangrene | |
|---|---|
| E1051 Dx angiopathy without gangrene ICD-10 E1052 Dx Type 1 diabetes mellitus with diabetic peripheral angiopathy with gangrene E1151 ICD-10 Dx Type 2 diabetes mellitus with diabetic peripheral angiopathy without gangrene ICD-10 Type 2 diabetes mellitus with diabetic peripheral angiopathy with gangrene E1152 Dx ICD-10 Other specified diabetes mellitus with diabetic peripheral angiopathy without gangrene ICD-10 Other specified diabetes mellitus with diabetic peripheral angiopathy without gangrene ICD-10 Other specified diabetes mellitus with diabetic peripheral angiopathy with gangrene ICD-10 Atherosclerosis of aorta | |
| E1052 Dx angiopathy with gangrene E1151 ICD-10 Dx Type 2 diabetes mellitus with diabetic peripheral angiopathy without gangrene ICD-10 Type 2 diabetes mellitus with diabetic peripheral angiopathy with gangrene E1152 Dx angiopathy with gangrene ICD-10 Other specified diabetes mellitus with diabetic peripheral angiopathy without gangrene ICD-10 Other specified diabetes mellitus with diabetic peripheral angiopathy with gangrene ICD-10 Other specified diabetes mellitus with diabetic peripheral angiopathy with gangrene ICD-10 Atherosclerosis of aorta | |
| ICD-10 Type 2 diabetes mellitus with diabetic peripheral angiopathy with gangrene E1152 Dx angiopathy with gangrene E1351 ICD-10 Other specified diabetes mellitus with diabetic peripheral angiopathy without gangrene ICD-10 Other specified diabetes mellitus with diabetic peripheral angiopathy without gangrene ICD-10 Other specified diabetes mellitus with diabetic peripheral angiopathy with gangrene ICD-10 Atherosclerosis of aorta | |
| E1152 Dx angiopathy with gangrene E1351 ICD-10 Other specified diabetes mellitus with diabetic peripheral angiopathy without gangrene ICD-10 Other specified diabetes mellitus with diabetic peripheral angiopathy with gangrene ICD-10 Dx Dx Atherosclerosis of aorta | |
| Dx peripheral angiopathy without gangrene ICD-10 Other specified diabetes mellitus with diabetic peripheral angiopathy with gangrene ICD-10 Dx Atherosclerosis of aorta | |
| E1352 Dx peripheral angiopathy with gangrene I700 ICD-10 Dx Atherosclerosis of aorta | |
| Dx Atherosclerosis of aorta | |
| 100.10 | |
| $\begin{array}{ c c c c c }\hline I701 & \begin{array}{ c c c c c }\hline ICD-10 \\ Dx \end{array} & \text{Atherosclerosis of renal artery} \end{array}$ | |
| I70201 ICD-10 Unspecified atherosclerosis of native arteries of extremities, right leg | |
| ICD-10 Unspecified atherosclerosis of native arteries of extremities, left leg | |
| ICD-10 Unspecified atherosclerosis of native arteries of extremities, bilateral legs | |
| ICD-10 Unspecified atherosclerosis of native arteries of extremities, other extremity | |
| ICD-10 Unspecified atherosclerosis of native arteries of extremities, unspecified extremity | |
| ICD-10 Atherosclerosis of native arteries of extremities with intermittent claudication, right leg | h |
| ICD-10 Atherosclerosis of native arteries of extremities with intermittent claudication, left leg | h |
| ICD-10 Atherosclerosis of native arteries of extremities with intermittent claudication, bilateral legs | h |
| I70218 ICD-10 Atherosclerosis of native arteries of extremities with intermittent claudication, other extremity | h |


001-

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


**NIS Protocol** 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


**NIS Protocol** 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


**NIS Protocol** 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


| of<br>ot<br>of<br>ot |
|----------------------|
| of<br>ver |
| of |
| of |
| of |
| of |
| of |
| of |
| of<br>er leg |
| of |
| of |
| of |
| of |
| of |
| of |
| of<br>remity |


**NIS Protocol** 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


**NIS Protocol** 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


| N055 ICD-10 Unspecified nephritic syndrome with diffuse mesangiocapillary glomerulonephritis ICD-10 Unspecified nephritic syndrome with dense department of the syndrome with dense department. | |
|---|---|
| ICD-10 Unspecified penbritic syndrome with dense der | |
| N056 Dx disease | posit |
| ICD-10 Unspecified nephritic syndrome with diffuse crescentic glomerulonephritis | |
| N058 ICD-10 Unspecified nephritic syndrome with other morphologic changes | |
| N059 ICD-10 Unspecified nephritic syndrome with unspecific morphologic changes | ed |
| N060 ICD-10 Isolated proteinuria with minor glomerular abnormality | |
| N061 ICD-10 Isolated proteinuria with focal and segmental glomerular lesions | |
| N062 ICD-10 Isolated proteinuria with diffuse membranous glomerulonephritis | |
| N063 ICD-10 Isolated proteinuria with diffuse mesangial proliferative glomerulonephritis | |
| N064 ICD-10 Isolated proteinuria with diffuse endocapillary proliferative glomerulonephritis | |
| N065 ICD-10 Isolated proteinuria with diffuse mesangiocapil glomerulonephritis | lary |
| N066 ICD-10 Isolated proteinuria with dense deposit disease | |
| N067 ICD-10 Isolated proteinuria with diffuse crescentic glomerulonephritis | |
| N068 ICD-10 Isolated proteinuria with other morphologic les | ion |
| N069 ICD-10 Isolated proteinuria with unspecified morpholo lesion | gic |
| N070 ICD-10 Hereditary nephropathy, not elsewhere classified with minor glomerular abnormality | ed |
| N071 ICD-10 Hereditary nephropathy, not elsewhere classified with focal and segmental glomerular lesions | ed |
| N072 ICD-10 Hereditary nephropathy, not elsewhere classified with diffuse membranous glomerulonephritis | ed |


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


001-

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


| m |
|---------|
| m right |
| m left |
| m |
| m right |
| m left |
| m |
| m |
| m right |
| m left |
| m other |
| m |
| ge |
| rain |

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


001-

**NIS Protocol**  Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


001-

**NIS Protocol**  Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| natic |
|--------------------|
| ed side |
| numatic<br>ninant |
| numatic<br>nant |
| numatic<br>- |
| numatic |
| numatic<br>ed side |
| natic<br>ninant |
| natic<br>nant |
| natic<br>- |
| natic |
| natic |
| natic<br>ed side |
| i |
| oid |


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


001-

**NIS Protocol** 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


001-

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies


# **BOEHRINGER INGELHEIM Group of Companies**

**NIS Protocol** 

c37262534-01 

| 99407 | СРТ | Smoking and tobacco use cessation counseling visit; intensive, greater than 10 minutes |
|---|---|---|
| 1032F | СРТ | Current tobacco smoker OR currently exposed to secondhand smoke (asthma) |
| 1033F | СРТ | Current tobacco nonsmoker AND not currently exposed to secondhand smoke (Asthma) |
| 1034F | СРТ | Current tobacco smoker (CAD, CAP, COPD, PV) (DM) |
| 1035F | СРТ | Current smokeless tobacco user (eg, chew, snuff) (PV) |
| 4000F | СРТ | Tobacco use cessation intervention, counseling (COPD, CAP, CAD, Asthma)(DM)(PV) |
| 4001F | СРТ | Tobacco use cessation intervention, pharmacologic therapy (COPD, CAP,CAD, Asthma)(DM)(PV) |

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### ANNEX 4. REVIEWERS AND APPROVAL SIGNATURES

The NIS Protocol must be sent for review to the following individuals prior to approval.

| Reviewer | NIS involving BI product(s) | NIS not involving BI product(s) | |
|---|---|---|---|
| | | Global<br>NIS | Local NIS |
| NIS Lead | X | X | X |
| Global TM Epi | X | X | X |
| Global TMM / TMMA / TM<br>Market Access | X | X | |
| Global Project Statistician | X | X | |
| Global TM RA | X | | |
| Global PVWG Chair | X | | |
| GPV SC | X | X | X |
| Global CTIS representative | X | | |
| Local Medical Director | X (if local study) | | X |
| Local Head MAcc / HEOR<br>Director | X (if local study) | | X |
| Global TA Head Epi* | X | X | |
| Global TA Head Clinical Development / Medical Affairs / Market Access* | X | X | |
| Global TA Head PV RM* | X | | |
| RWE CoE | X | X | |
| PSTAT / PSTAT-MA<br>(for NISnd only) | X | X | X |
| NIS DM | X | X | X |
| Local Head MA/Clinical<br>Development | | | X (does not apply to<br>NISed without chart<br>abstraction) |

<sup>\*</sup> After review by Global TM for function

Stiolto vs Trelegy V1.0 04 May



#### APPROVAL / SIGNATURE PAGE

Document Number: c37262534 Technical Version Number: 1.0

**Document Name:** nis-us-heor-stiolto-vs-trelegy-study-protocol

**Title:** Health Care Resource Utilization, Cost and Other Outcomes of Patients Diagnosed with COPD Initiating Tiotropium Bromide/Olodaterol versus Fluticasone Furoate/Umeclidinium/Vilanterol

## **Signatures (obtained electronically)**

| Meaning of Signature | Signed by | Date Signed |
|----------------------|-----------|------------------------|
| Approval | | 31 Mar 2022 15:44 CEST |
| Approval | | 31 Mar 2022 15:52 CEST |
| Approval | | 31 Mar 2022 16:54 CEST |

Boehringer IngelheimPage 2 of 2Document Number: c37262534Technical Version Number:1.0

## (Continued) Signatures (obtained electronically)

| Meaning of Signature Signed by Date Signed |
|--------------------------------------------|
|--------------------------------------------|